CLINICAL TRIAL: NCT01135056
Title: Phase III Multi-Centre Open-Label Randomized Controlled Trial of Selective Internal Radiation Therapy (SIRT) Versus Sorafenib in Locally Advanced Hepatocellular Carcinoma (SIRveNIB)
Brief Title: Study to Compare Selective Internal Radiation Therapy (SIRT) Versus Sorafenib in Locally Advanced Hepatocellular Carcinoma (HCC)
Acronym: SIRveNIB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: National Cancer Centre, Singapore (Other); National Medical Research Council (NMRC), Singapore (Other Government); Singapore Clinical Research Institute (Other); Sirtex Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHCC06
Record Dates: First submitted 2010-05-24; First posted 2010-06-02 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Randomized; Open-label; Multi-Centre; Phase III; Sorafenib; SIR-Spheres
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib, Multikinase Inhibitor, Tablet (Active Comparator): Sorafenib tosylate:
  Sorafenib is a multikinase inhibitor that decreases tumor cell proliferation.
  Sorafenib was shown to inhibit multiple intracellular (c-CRAF, BRAF and mutant BRAF) and cell surface kinases (KIT, FLT- 3, RET, VEGFR-1, VEGFR- 2, VEGFR- 3, and PDGFR- ß). Several of these kinases are thought to be involved in tumor cell signaling, angiogenesis and apoptosis. Sorafenib inhibited tumor growth of the human hepatocellular carcinoma and renal cell carcinoma, and several other human tumor xenografts in immunocompromised mice. A reduction in tumor angiogenesis and increases in tumor apoptosis was seen in models of human hepatocellular and renal cell carcinoma. Additionally a reduction in tumor cell signaling was seen in a model of human hepatocellular carcinoma.
  Interventions: Drug: Sorafenib tosylate
- SIR-Spheres, Microspheres, Device (Active Comparator): SIR-Spheres:
  SIR-Spheres consist of biocompatible resin microspheres containing yttrium-90, with a size between 20 and 60 microns in diameter. Yttrium-90 is a high-energy pure beta-emitting isotope with no primary gamma emission. The half life of yttrium-90 is 64.1 hours. In clinical use which requires the isotope to decay to infinity, 94% of the radiation is delivered in 11 days leaving only background radiation with no therapeutic value.
  SIR-Spheres is implanted into hepatic tumours by delivery via either the common hepatic artery or the right or left hepatic artery using a catheter or implanted port . Once SIR-Spheres is implanted into the liver, it is not metabolised or excreted and it stays permanently in the liver.
  Interventions: Device: SIR-Spheres

INTERVENTIONS:
Device: SIR-Spheres — One time treatment. Dose administered based on tumour volume. Each vial is 3.0GBq.
  Other Names: Yttrium-90 Microspheres
  Arms: SIR-Spheres, Microspheres, Device
Drug: Sorafenib tosylate — Oral Tablet, 400mg B.i.d, until progression or unacceptable toxicity develops
  Other Names: Nexavar
  Arms: Sorafenib, Multikinase Inhibitor, Tablet

SUMMARY:
The primary objective of this study is to assess the efficacy of SIRT as compared with Sorafenib in patients with locally advanced liver cancer in terms of overall survival (OS).

The Study null hypothesis is, there is no difference in overall survival between patients receiving SIRT and those receiving Sorafenib therapy.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the 5th most common cancer worldwide but unfortunately between 70 - 80% of all HCC are in the Asia-Pacific because of the prevalence of chronic viral hepatitis in the region. The increase in the prevalence of chronic hepatitis C in the Western world however predicts that HCC will similarly be an important cause of death there in the next 20 years.

Only 15-20% of HCC are today potentially curable by surgery at the time of diagnosis. Another 10-15% of patients may benefit from potentially curative locally ablative therapy such as radio-frequency ablation. Prognosis in the majority of patients has been dismal as conventional systemic therapies have been largely inefficacious. The first successfully trialed systemic targeted therapy, sorafenib (2007) prolonged survival by a modest average of 3 months in patients with good underlying liver function.

While the liver is radio-sensitive, external beam radiation causes significant radio-toxicity. To overcome this, selective internal radiation therapy (SIRT) was developed to deliver a radiation source directly to liver cancer via the arterial route. Sir-sphere is radioactive yttrium on a 90 micro-meter diameter resin carrier and is an established therapy in colorectal metastasis. Sir-sphere has been reported to cause significantly tumour regression in HCC.

This study will evaluate the efficacy of SIRT using SIR-Spheres yttrium-90 microspheres compared to sorafenib in the treatment of patients with locally advanced primary HCC.

ELIGIBILITY:
Inclusion Criteria:

* Disease must be locally advanced as defined by BCLC (B) intermediate stage or BCLC (C) advanced stage without extra-hepatic disease (only with branch portal vein thrombosis).
* Willing, able and mentally competent to provide written informed consent prior to any testing undertaken for this study protocol, including screening tests and evaluations that are not considered to be part of the subject's routine care.
* Aged 18 years/older (either gender).
* Unequivocal diagnosis of HCC.
* HCC not amenable to surgical resection or immediate liver transplantation, or cannot be optimally treated with local ablative techniques such as RFA, consistent with the practice of the clinical trial centre.
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with spiral CT scan or MRI.
* ECOG performance status 0-1.
* Child-Pugh A-B (up to 7 points)
* Adequate haematological, renal and hepatic function as follows:
* Leukocytes ≥ 2,500/μL
* Platelets ≥ 80,000/μL
* Haemoglobin > 9.5g/dL
* Total bilirubin < 2.0mg/dL
* INR ≤ 2.0
* ALP ≤ 5 x institutional ULN
* AST and ALT ≤ 5 x institutional ULN
* Albumin ≥ 2.5g/dL
* Creatinine ≤ 2.0mg/dL
* Life expectancy of at least 3 months without any active treatment.
* Suitable for protocol treatment as determined by clinical assessment undertaken by the Investigator.
* Female patients must be either postmenopausal or, if premenopausal, must have a negative pregnancy test and agree to use 2 forms of contraception if sexually active during their study participation.
* Male patients must be surgically sterile, or if sexually active and having a pre-menopausal female partner then must be using an acceptable form of contraception.

Exclusion Criteria:

* Have had more than 2 administrations of hepatic artery directed therapy.
* Subjects who have had hepatic artery directed therapy done < 4 weeks prior to study entry.
* Have had systemic chemotherapy for HCC except for prior adjuvant or neoadjuvant therapy given more than 6 months from enrolment.
* have had prior treatment with Sorafenib or VEGF inhibitors.
* Prior hepatic radiation therapy for HCC or other malignancy.
* Currently receiving any other investigational agents for the treatment of their cancer.
* Has intractable clinical ascites (in spite of optimal diuretic treatment) or any other clinical signs of liver failure, on physical examination.
* Complete main portal vein thrombosis.
* Any metastatic disease (local-regional lymph nodes measuring less than 2 cm in greatest diameter or lung nodules measuring less than 1 cm are not contraindications as per Investigator discretion).
* Any other concurrent malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least 5 years.
* Presence of clinical signs of CNS metastases due to their poor prognosis and because progressive neurologic dysfunction would confound the evaluation of neurologic and other adverse events.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection (except viral hepatitis), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any of the following contraindications to angiography and selective visceral catheterization:
* Bleeding diathesis, not correctable by the standard forms of therapy.
* Severe peripheral vascular disease that would preclude arterial catheterization.
* Portal hypertension with hepato-fugal flow as documented on baseline spiral CT scan.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SIR-Spheres or Sorafenib.
* Inability or unwillingness to understand or sign a written informed consent document.
* Female subjects who are pregnant or currently breastfeeding.
* Female subjects, unless postmenopausal or surgically sterile, unwillingness to practice effective contraception, as per Investigator discretion during the study. The rhythm method is not to be used as the sole method of contraception.
* Male subjects, unwillingness to practice effective contraception (per Investigator discretion) while taking part in this study, because the effect of the SIR-Spheres treatment on sperm or upon the development of an unborn child are unknown.
* Current enrolment in any other investigational therapeutic drug or device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2010-07; Primary Completion 2018-07-31 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2 years
  Overall Survival is defined as the time from the date of randomisation to the date of death due to any cause. All patients will be followed up until death to compare the overall survival between the two treatments. 2 years is an estimated time frame.

SECONDARY OUTCOMES:
Progression free survival in the liver | 2 years
  Progression-free survival in the liver is defined as the time interval between randomisation and the date of tumour progression in the liver or death, whichever is earlier. Tumour progression in the liver will be determined from serial CT scans. Diagnosis of tumour progression of disease should be made using the RECIST guideline version 1.1. 2 years is an estimated time frame.
Progression free survival overall | 2 years
  Progression-free survival overall is defined as the time interval between randomisation and the date of tumour progression at any site in the body or death, whichever is earlier. Tumour progression at any site in the body will be measured by any definitive imaging technique including CT scan, MRI study or other nuclear medicine scan. The Investigator should clearly indicate the site of tumour progression (hepatic or extra-hepatic) at the time of recurrence.
  2 years is an estimated time frame.
Tumour Response Rate | 2 years
  Tumour response and progression will be evaluated in this study using the new response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1) [European Journal of Cancer (45): 228 - 247, 2009] (http://ctep.cancer.gov/protocolDevelopment/docs/recist_guideline.pdf).
  2 years is an estimated time frame
Toxicity and Safety | Up to 2 years
  Toxicity will be assessed using the National Cancer Institute Common Terminology Criteria (NCI-CTC) version 4.02. Patients for both treatment arms will be followed-up for safety and toxicity from the time of study entry (randomisation day) until 30 days post study conclusion or until commencement of the next alternative therapy, which ever is earlier.
Health Related Quality of Life (QoL) | Up to 2 years
  Quality of life (QoL) will be measured by using the EQ-5D questionnaire over the study period. QoL for patients will be measured until their first disease progression up to 2 years (estimated) which ever is earlier.
Liver resection rate | Up to 2 years
  Patients will be assessed for suitability for liver resection every 12 weekly until their study conclusion up to 2 years which ever is earlier.
Liver Transplantation Rate | Up to 2 years
  Patients will be assessed for suitability for liver transplantation every 12 weekly until their study conclusion up to 2 years which ever is earlier.
Time to Disease Progression | Up to 2 years
  Time to Disease Progression (TTP) is defined as a measure of time after a disease is diagnosed (or treated) until the disease starts to get worse. Disease Progression will be measured by RECIST guideline version 1.1. TTP will be measured every 12 weekly up to 2 years (estimated).
Disease control rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierce KH Chow, MBBS, PhD, Study Chair — National Cancer Centre, Singapore
Locations (29):
- The Brunei Cancer Centre, Kampong Jerudong, Brunei, Brunei
- Yangon GI & Liver Centre, Yangon, Burma
- Queen Mary Hospital, Hong Kong, Hong Kong, China
- Indonesia (2):
  - University of Udayana, Rumah Sakit Sanglah, Indonesia, Denpasar, Bali
  - Cipto Mangunkusumo Hospital ,University of Indonesia, Jakarta
- Malaysia (3):
  - Penang Adventist Hospital, George Town, Pulau Pinang
  - Sarawak General Hospital, Kuching, Sarawak
  - University Malaya Medical Center, Kuala Lumpur
- National Cancer Center of Mongolia, Ulaanbaatar, Mongolia
- Auckland City Hospital, Grafton, Auckland, New Zealand
- Philippines (4):
  - Makati Medical Center, Manila, Makati City
  - The Medical City, Pasig, Manila
  - St. Luke's Medical Center, Philippines, Quezon City, Manila
  - Davao Doctors Hospital, Davao City
- Singapore (4):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - National Cancer Center Singapore, Singapore
  - Khoo Teck Puat Hospital, Singapore
- South Korea (5):
  - Severance Hospital, Yonsei University College of Medicine, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul
- Taiwan (5):
  - National Taiwan University Hospital, Taipei City, Taipei
  - Taipei Veterans General Hospital, Taipei City, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District, Taoyuan Hsien
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
- Chulabhorn Hospital, Bangkok, Thailand

REFERENCES:
- [Derived] Chow PKH, Gandhi M, Tan SB, Khin MW, Khasbazar A, Ong J, Choo SP, Cheow PC, Chotipanich C, Lim K, Lesmana LA, Manuaba TW, Yoong BK, Raj A, Law CS, Cua IHY, Lobo RR, Teh CSC, Kim YH, Jong YW, Han HS, Bae SH, Yoon HK, Lee RC, Hung CF, Peng CY, Liang PC, Bartlett A, Kok KYY, Thng CH, Low AS, Goh ASW, Tay KH, Lo RHG, Goh BKP, Ng DCE, Lekurwale G, Liew WM, Gebski V, Mak KSW, Soo KC; Asia-Pacific Hepatocellular Carcinoma Trials Group. SIRveNIB: Selective Internal Radiation Therapy Versus Sorafenib in Asia-Pacific Patients With Hepatocellular Carcinoma. J Clin Oncol. 2018 Jul 1;36(19):1913-1921. doi: 10.1200/JCO.2017.76.0892. Epub 2018 Mar 2. PMID 29498924
- [Derived] Gandhi M, Choo SP, Thng CH, Tan SB, Low AS, Cheow PC, Goh AS, Tay KH, Lo RH, Goh BK, Wong JS, Ng DC, Soo KC, Liew WM, Chow PK; Asia-Pacific Hepatocellular Carcinoma Trials Group. Single administration of Selective Internal Radiation Therapy versus continuous treatment with sorafeNIB in locally advanced hepatocellular carcinoma (SIRveNIB): study protocol for a phase iii randomized controlled trial. BMC Cancer. 2016 Nov 7;16(1):856. doi: 10.1186/s12885-016-2868-y. PMID 27821083
- See also: AHCC Trials Group — http://www.scri.edu.sg/crn/asia-pacific-hepatocellular-carcinoma-ahcc-trials-group/about-ahcc/